CLINICAL TRIAL: NCT05569798
Title: Acceptability and Feasibility of Interprofessional Scheduled Whole-Body Point-of-Care Ultrasound in the Intensive Care Unit: A Randomised Controlled Feasibility Trial
Brief Title: The INSIGHT Feasibility Study Ultrasound in the Intensive Care Unit: A Randomised Controlled Feasibility Trial
Acronym: INSIGHT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 313425
Record Dates: First submitted 2022-09-27; First posted 2022-10-06 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Cardiac Complication; Pleural Effusion; Consolidation; Ascites; Thrombosis
MeSH Terms: conditions — Critical Illness; Pleural Effusion; Ascites; Thrombosis

STUDY DESIGN:
Intervention Model Description: A parallel single centre feasibility randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Thirty patients will receive standard care (regular ICU treatment without any restriction to usual medical care). INSIGHT scans will not be performed on these patients. However, other forms of ultrasound scanning will be permitted in this group. For example, departmental ultrasound scans (full echocardiography, liver, or vascular ultrasound assessment); transoesophageal echocardiography; transcranial doppler; any form of PoCUS other than the INSIGHT scan.
- Standard care + the INSIGHT intervention (Experimental): Thirty patients will receive standard care + the INSIGHT intervention. The INSIGHT intervention is described in detail in section 5.7.1. INSIGHT scans will be performed by staff trained in the INSIGHT Training and Competency Programme on days 1 (0-36 hours), 3 (72-96 hours) and 7 (6 to 8 days) from ICU admission. Scans will only be performed at these timepoints if the patient is still admitted to the ICU.
  Interventions: Diagnostic Test: Whole body point of care ultrasound scan

INTERVENTIONS:
Diagnostic Test: Whole body point of care ultrasound scan — The INSIGHT Scan is a whole-body PoCUS scan which comprises imaging the following windows:
  1. subcostal
  2. inferior vena cava cardiac view
  3. left hemidiaphragm
  4. bladder
  5. right hemidiaphragm
  6. six major central veins (left/right internal jugular/ subclavian/ femoral veins)
  The scan should take no more than 10 minutes to perform. Simple yes/no questions are asked for each window to identify any significant abnormalities. For example, is the left ventricle bigger than the right ventricle; is there a pleural effusion; is the bladder distended etc.
  The scan is reported in the intensive care online medical notes and reviewed by the clinical team as soon as possible.
  Other Names: The INSIGHT scan
  Arms: Standard care + the INSIGHT intervention

SUMMARY:
Point-of-care ultrasound (PoCUS) is a rapidly evolving method of clinical assessment within the intensive care unit (ICU) with training predominantly aimed at physicians. Routine whole-body PoCUS (lungs, heart, abdomen and blood vessels) when conducted by physicians benefits patient care and outcomes including reducing the risk of prolonged ICU stay (>7 days) and mechanical ventilation as well as reducing utilisation of other diagnostic tests. However, physician-only use of PoCUS does not allow for use as a routine assessment method in the ICU due to the low physician to patient ratio and poor ultrasound accreditation rate.

Providing other healthcare professionals such as Advanced Critical Care Practitioners (ACCPs), ICU nurses and physiotherapists with PoCUS skills increases the proportion of trained staff to perform routine PoCUS in the ICU. This could aid earlier identification of abnormal pathology, earlier treatment, and prevent patient deterioration. The advancement of handheld PoCUS technology is making ultrasound more portable, cheaper and easier to use.

The increased accessibility of PoCUS combined with growing evidence of its diagnostic accuracy compared to other modes of imaging means PoCUS use is gaining traction globally. However, little to no research exists investigating the feasibility of implementing scheduled interprofessional PoCUS in the ICU and its impact on patient outcomes.

This study aims to evaluate the acceptability and feasibility of a quick and simple whole body ultrasound scan performed by trained ACCPs, ICU nurses, physiotherapists, and doctors at set time points throughout the patients ICU stay. The investigators want to find out the most common barriers and facilitators to intervention implementation and to explore the key clinical outcomes for use in a future definitive RCT.

DETAILED DESCRIPTION:
PoCUS is a non-invasive procedure that does not use harmful radiation. PoCUS therefore minimises patient risk and has superior diagnostic capabilities compared to the stethoscope. Non-medics can learn and utilise PoCUS with comparable accuracy. Routine whole-body PoCUS could enable more informed and timely clinical decision-making regarding lifesaving interventions such as patient positioning (proning), ventilatory support, and fluid balance optimisation. PoCUS could decrease time spent in diagnostic testing outside the ICU, minimising spread of infection through reduced patient contact, and reduce risk associated with patient transfers to scanning. Increased PoCUS use therefore has the potential to positively impact more patients, with less disruption to patient care.

In addition, increased routine PoCUS use by multiple professions will create a shared communication platform with the potential to enhance interdisciplinary collaboration. PoCUS use meets the growing demand for advanced assessment skills in the ICU, increasing autonomy and improving staff retention. PoCUS may reduce service costs by limiting the need for other imaging. In addition, the economic value of fewer diagnostic tests and the potential for improved patient outcomes could be significant. Storage solutions for diagnostic imaging present an ongoing challenge throughout the healthcare service. Imaging is stored on multiple platforms, making reviewing of images often location dependent. Identifying the most accessible storage platform for routine image review could significantly influence utilisation of images during patient assessment.

The investigator's aim is to evaluate the acceptability and feasibility of the INSIGHT Intervention within the ICU environment. This comprises performing a whole body PoCUS (INSIGHT) scan on days 1, 3, and 7 of ICU admission, with review by the clinical team.

The INSIGHT Scan is a whole-body PoCUS scan which comprises imaging the following windows:

1. subcostal
2. inferior vena cava cardiac view
3. left hemidiaphragm
4. bladder
5. right hemidiaphragm
6. six major central veins (left/right internal jugular/ subclavian/ femoral veins)

Design and Setting: A mixed-methods study across 2 adult ICUs (30 beds) within the critical care centre at KCH, London.

The Study will be conducted in two stages:

Stage 1 Aim: The aim of this stage is to identify and address the acceptability and feasibility of the INSIGHT intervention from the perspective of key stakeholders.

The primary objectives will be to:

1. Assess barriers and facilitators to delivering the delivering the INSIGHT intervention
2. Refine the INSIGHT intervention so that it is acceptable to key stakeholders
3. To have a clear understanding of intervention fidelity and ability to recruit participants (33, 34)

The following feasibility outcomes will be evaluated:

1. availability of a trained staff member to perform the INSIGHT scan when an eligible patient is identified
2. barriers to completing the INSIGHT scan
3. barriers to accessing INSIGHT scan images during ward round
4. barriers to incorporating the INSIGHT scan into routine clinical care
5. number of eligible patients (screening data)
6. screening and recruitment methods (number of 'missed' patients and reason for non-enrolment)

ICU Patient Sample: Convenience sampling will be used to recruit 20 adult (18 years or over) ICU patients.

ICU Staff Sample: Prior to stage 1 commencement, a minimum of 10 staff members will have completed the training and will be approached for consent to participate in this study.

Fifteen INSIGHT-trained and non INSIGHT-trained clinical staff will be recruited using purposive sampling (ACCPs, nurses, doctors, physiotherapists) to either attend one of two focus groups.

Data collection methods:

* Go-along interviews with trained staff whilst performing the INSIGHT scan
* Ward round observations
* Questionnaires will be distributed to staff before any patients receive an INSIGHT scan, the after 5, 10, 15, and 20 patients have been scanned
* Focus groups

Stage 2 Aim: To evaluate the feasibility of the INSIGHT intervention trial design to inform a future adequately powered randomised controlled trial.

Primary Objective: To evaluate the feasibility of a randomised controlled trial of the INSIGHT Scanning Protocol.

Feasibility objectives:

1. Recruitment rate and willingness of approached eligible patients to consent
2. Number of complete scans (i.e., 6/6 windows)
3. Reasons scans not performed/completed
4. Time taken to perform and report INSIGHT scans
5. Proportion of complete scan reports compared to the total number of scans performed
6. Staff perceived feasibility of the INSIGHT Scan on days 1, 3, and 7 of ICU admission

6. Adherence to the INSIGHT Scanning Protocol, measured by the number of INSIGHT scans and reports completed compared to the number required in the INSIGHT protocol design 7. Rate of adverse and serious adverse events

Exploratory clinical objectives:

1. Number of diagnostic tests (chest X-ray, non-INSIGHT ultrasound, CT scans [excluding head]) per patient during ICU stay
2. Radiation exposure (measured in mSv)
3. Duration of mechanical ventilation
4. ICU length of stay
5. Number of nosocomial infections
6. Number and type of incidental clinical findings detected using the INSIGHT scan and time to a clinical intervention to address this incidental clinical finding

Patient participant sample: The investigators will recruit 60 patients during the study.

Randomisation: Participants will be randomised to receive the INSIGHT intervention or standard care (no INSIGHT intervention) on a 1:1 basis.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Patients 18 years of age or more
2. Critically ill patient requiring level 2/3 care
3. Provides consent to participate (or consent given by substitute decision maker)
4. Anticipated to be admitted to ICU for at least 72 hours from time of admission

Patient Exclusion Criteria:

1. Injuries that prevent probe positioning:

   1. Dressings that restrict the INSIGHT window views
   2. Flail chest
   3. Other unstable fractures that might prevent scanning
   4. Open abdominal/thorax wounds
   5. Surgical emphysema
2. Uncontrolled agitation or pain: this will make scanning more challenging and affect image acquisition
3. Clinical instability requiring prioritisation of stabilising or resuscitative care
4. Allergy to ultrasound gel
5. Anticipated withdrawal of care in the next 24 hours

Staff Inclusion Criteria

i. Nurse, ACCP, physiotherapist, or doctor ii. Completion of an advanced course in ICU nursing, ACCP course, ICU physiotherapy or medicine iii. Working in a participating ICU for a minimum of 6 months before enrolment on training course iv. Competent or undergoing training in the INSIGHT Scan

ICU staff exclusion criteria

i. Any injuries or musculoskeletal conditions that would be exacerbated by performing ultrasound ii. On rotation or planning on leaving ICU role in 6 or less months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-12-04 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Adherence to the INSIGHT Scanning Protocol, measured by the number of INSIGHT scan reports completed compared to the number required in the INSIGHT protocol design | Day of ICU admission (day 1) to day 7 of ICU admission
  Scanning timepoints are on days 1, 3, and 7 of ICU admission. However the patient may have been discharged before the second or third timepoint. This measure therefore captures feasibility of performing the scan during the available opportunities only.
Recruitment rate and willingness of approached eligible patients to consent | Through to study completion, approximately 18 months
  We will capture those who do not consent in a screening log
Number of complete scans (i.e., 6/6 windows) | Through to study completion, approximately 18 months
  The proportion of ultrasound scans that are completed
Reasons scans not performed/completed | Through to study completion, approximately 18 months
  We will capture reasons for not completing scan in the ultrasound report
Proportion of complete scan reports compared to the total number of scans performed | Through to study completion, approximately 18 months
Staff perceived feasibility of the INSIGHT Scan on days 1, 3, and 7 of ICU admission | 18 months
  We will capture this during semi-structured 30 minute interviews
Rate of adverse and serious adverse events | Through to study completion, approximately 18 months

OTHER OUTCOMES:
Number of diagnostic tests (chest X-ray, non-INSIGHT ultrasound, CT scans [excluding head]) per patient during ICU stay | Day of ICU admission to day 28 or ICU discharge/death
Radiation exposure | Day of ICU admission to day 28 or ICU discharge/death
  measured in millisievert
Duration of mechanical ventilation | Day of ICU admission to day 28 or ICU discharge/death
  Multiple episodes will be recorded if patient is reintubated
ICU length of stay | Day of ICU admission to day 28 or ICU discharge/death
Number and type of nosocomial infections | Day of ICU admission to day 28 or ICU discharge/death
  site of infection, organism confirmed by microbiology, antibiotic treatment, date started, date stopped will all be collected
Number and type of incidental clinical findings detected using the INSIGHT scan | Day of ICU admission (day 1), day 3, and day 7 of ICU admission
  Findings include: Pericardial effusion; Dilated right ventricle; Abnormal contractility and function of the left or right ventricle; Lung consolidation; Pleural effusion; Presence of 3 or more B-lines; Abdominal fluid collection; Abnormal growth/ thrombus in any view
Time from ICU admission (or from INSIGHT scan if performed on days 3 and 7) to clinical | Day of ICU admission to day 28 or ICU discharge/death
  Interventions include: Insertion of central venous catheter; Commencement of first vasopressors whilst in ICU; Renal filtration; Start of first antibiotics prescribed in ICU; Drain inserted (specify type); ECG; Insertion of urinary catheter; Repositioning of existing urinary catheter; Other (please specify)

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Corcoran, Principal Investigator — Doctoral Research Fellow
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
The data collected will only be used for publications relating to this trial. Relevant data to the publications will be published. More detailed datasets will be available on request. However these data cannot be used for any other research.